CLINICAL TRIAL: NCT05362058
Title: A Phase 3, Parallel-Design, Open-Label, Randomized Control Study to Evaluate the Efficacy and Safety of LY3209590 as a Weekly Basal Insulin Compared to Insulin Degludec in Insulin Naïve Adults With Type 2 Diabetes
Brief Title: A Study of Insulin Efsitora Alfa (LY3209590) Compared to Degludec in Adults With Type 2 Diabetes Who Are Starting Basal Insulin for the First Time
Acronym: QWINT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18262; I8H-MC-BDCX (Other: Eli Lilly and Company); 2021-005891-21 (EudraCT Number)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 500 U/mL - Insulin Efsitora Alfa (Experimental): * Participants received 500 units per milliliter (U/mL) of insulin efsitora alfa administered subcutaneously (SC) once weekly (QW) over a 52-week treatment period, followed by a 5-week safety follow-up period.
  * Participants continued their protocol-specified stable therapy with non-insulin antihyperglycemic medications throughout the study, at the discretion of the investigator.
  Interventions: Drug: Insulin Efsitora Alfa
- 100 U/mL - Insulin Degludec (Active Comparator): * Participants received 100 U/mL insulin degludec administered SC once daily (QD) over a 52-week treatment period, followed by a 5-week safety follow-up period.
  * Participants continued their protocol-specified stable therapy with non-insulin antihyperglycemic medications throughout the study, at the discretion of the investigator.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Insulin Efsitora Alfa — Administered SC
  Other Names: LY3209590 and Basal Insulin-FC
  Arms: 500 U/mL - Insulin Efsitora Alfa
Drug: Insulin Degludec — Administered SC
  Arms: 100 U/mL - Insulin Degludec

SUMMARY:
The purpose of this study is to determine the effect and safety of insulin efsitora alfa (LY3209590) compared to degludec in adult participants with type 2 diabetes who are starting basal insulin for the first time. The study consists of a 1-week screening period, a 2-week lead-in period, a 52-week treatment period, and a 5-week safety follow-up period. The study will last up to 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of Type 2 diabetes (T2D) according to the World Health Organization Criteria
* Have an Hemoglobin A1c (HbA1c) of 7.0 percent (%) - 10.5% inclusive, at screening
* Are on a stable treatment with 1 to 3 antihyperglycemic medication for at least 3 months prior to screening and willing to continue the stable treatment for the duration of the study
* These antihyperglycemic medications are accepted in the study

  * dipeptidyl peptidase-4 (DPP-4) inhibitors
  * sodium-glucose cotransporter 2 (SGLT2) inhibitors
  * biguanides, such as metformin
  * alpha-glucosidase inhibitors
  * glucagon-like peptide-1 (GLP-1) receptor agonists, oral or injectable
  * Sulfonylureas, or
  * Thiazolidinediones.
* Are insulin naïve.

Exceptions:

* short-term insulin treatment for a maximum of 14 days, prior to screening, and prior insulin treatment for gestational diabetes

  * Have a body mass index of less than or equal to (≤) 45 kilogram/square meter (kg/m²).

Exclusion Criteria:

* Have a diagnosis of Type 1 diabetes (T1D), latent autoimmune diabetes, or a specific type of diabetes other than T2D, for example, monogenic diabetes, diseases of the exocrine pancreas, or drug-induced or chemical-induced diabetes.
* Have a history of greater than (>) 1 episode of ketoacidosis or hyperosmolar state or coma requiring hospitalization within 6 months prior to screening. Have had severe hypoglycemia episodes within 6 months prior to screening. Have a history of renal transplantation, are currently receiving renal dialysis, or have an estimated glomerular filtration rate.
* Have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c.
* Have had New York Heart Association Class IV heart failure or any of these cardiovascular conditions within 3 months prior to screening

  * Acute myocardial infarction
  * Cerebrovascular accident (stroke), or
  * Coronary bypass surgery.
  * Have had gastric bypass (bariatric) surgery, restrictive bariatric surgery, for example Lap-Band, or sleeve gastrectomy within 1 year prior to screening
  * Have had significant weight gain or loss within 3 months prior to screening, for example, greater than or equal to (≥) 5%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (113):
- United States (30):
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Valley Research, Fresno, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - Catalina Research Institute, LLC, Montclair, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - New West Physicians Clinical Research, Golden, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - East Coast Institute for Research - Canton, Canton, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Qualmedica Research, Bowling Green, Kentucky
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - SKY Clinical Research Network Group-Quinn, Ridgeland, Mississippi
  - Clinvest Research LLC, Springfield, Missouri
  - Clarity Clinical Research, East Syracuse, New York
  - Great Lakes Medical Research, LLC, Westfield, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Intend Research, LLC, Norman, Oklahoma
  - Jefferson Clinical Research Institute (JCRI), Philadelphia, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Multicare Institute for Research and Innovation, Spokane, Washington
- Brazil (7):
  - CEDOES, Vitória, Espírito Santo
  - Cline Research Center, Curitiba, Paraná
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Hospital São Lucas de Copacabana, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Canada (7):
  - LMC Diabetes & Endocrinology, Brampton, Ontario
  - Aggarwal and Associates Limited, Brampton, Ontario
  - LMC Manna Research, Ottawa, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Centricity Research Etobicoke Endocrinology, Toronto, Ontario
  - Fadia El Boreky Medicine, Waterloo, Ontario
  - 9109-0126 Quebec Inc., Montreal, Quebec
- China (26):
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Hebei Medical University - Harrison International Peace Hospital, Hengshui Shi, Hebei
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Jiangyin Hospital of Southeast University Medical College, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Putuo District Center Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Zhu Xianyi Memorial Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
- Czechia (7):
  - INTENDIA klinika s.r.o., Chrudim III, Chrudim
  - MUDr. Alena Vachova, České Budějovice, Jihočeský kraj
  - MUDr. Tomas Edelsberger, Krnov, Moravskoslezský kraj
  - Diahelp s.r.o, Pardubice V, Pardubice
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague, Praha 4
  - Diacentrum Brandys n.L. s.r.o., Brandýs nad Labem, Praha-vých
  - MUDr. Tomas Hrdina, Opočno, Rychnov Nad Kněžnou
- Germany (8):
  - Praxis Sauter & Sauter & Vorbach, Wangen, Baden-Wurttemberg
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - Diabetologikum Ludwigshafen/Die Praxis am Ludwigsplatz, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabeteszentrum Hamburg West, Hamburg
- Greece (4):
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro, Attikí (Region)
  - Alexandra Hospital, Athens, Attikí
  - Thermi Clinic, Thessaloniki, Thessaloníki
  - Athens Euroclinic, Athens
- Japan (18):
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya, Aichi-ken
  - Kashiwa City Hospital, Kashiwa, Chiba
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Nippon Kokan Fukuyama Hospital, Fukuyama-shi, Hiroshima
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - Manda Memorial Hospital, Sapporo, Hokkaido
  - MinamiAkatsukaClinic, Mito, Ibaraki
  - Nakakinen clinic, Naka, Ibaraki
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki, Kanagawa
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Shimizu Clinic Fusa, Saitama-shi, Saitama
  - Kumanomae Nishimura Clinic, Arakawa-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Hachioji Diabetes Clinic, Hachioji-shi, Tokyo
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - Tomonaga Clinic, Shinjuku, Tokyo
  - Yoshimura Clinic, Kumamoto
  - Abe Clinic, Ōita
- Investigacion En Salud Y Metabolismo Sc, Chihuahua City, Mexico
- Puerto Rico (2):
  - Centro de Endocrinologia y Nutricion, Caguas
  - Private Practice - Dr. Paola Mansilla-Letelier, Guaynabo
- South Korea (3):
  - Kangwon National University Hospital, Chuncheon, Kang-won-do
  - Hanyang University Guri Hospital, Guri-si, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teuk

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Miller E, Davidson MB, Bajaj HS, Rosenstock J, Philis-Tsimikis A, Bergenstal RM, Case M, Ilag L, Threlkeld R, Levasseur E, Gelsey F. Evaluation of Overall Health State, Treatment Burden, and Satisfaction with Insulin Efsitora Alfa (Efsitora) vs. Daily Comparator in Adults with Type 2 Diabetes in the QWINT Clinical Trial Program. Diabetes Ther. 2026 Jan 27. doi: 10.1007/s13300-025-01833-5. Online ahead of print. PMID 41591636
- [Derived] Wysham C, Bajaj HS, Del Prato S, Franco DR, Kiyosue A, Dahl D, Zhou C, Carr MC, Case M, Firmino Goncalves L; QWINT-2 Investigators. Insulin Efsitora versus Degludec in Type 2 Diabetes without Previous Insulin Treatment. N Engl J Med. 2024 Dec 12;391(23):2201-2211. doi: 10.1056/NEJMoa2403953. Epub 2024 Sep 10. PMID 39254740
- See also: A Study of LY3209590 Compared to Degludec in Adults With Type 2 Diabetes Who Are Starting Basal Insulin for the First Time (QWINT-2) — https://trials.lilly.com/en-US/find/completed?trialname=%20I8H-MC-BDCX&externalRequestID=68cbce79-fbf1-46c5-852a-338ca6e2be85

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants continued their protocol-specified stable therapy with 1 to 3 non-insulin antihyperglycemic medications, including glucagon-like peptide-1 receptor agonists (GLP-1 RA), as well as non-GLP-1 receptor agonists such as dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose cotransporter 2 (SGLT2) inhibitors, biguanides (e.g., metformin), alpha-glucosidase inhibitors, sulfonylureas (SUs), or thiazolidinediones throughout the study, at the discretion of the investigator.
Groups:
- 500 U/mL - Insulin Efsitora Alfa: - Participants received 500 units per milliliter (U/mL) of insulin efsitora alfa administered subcutaneously (SC) once weekly (QW) over a 52-week treatment period, followed by a 5-week safety follow-up period.
- 100 U/mL - Insulin Degludec: - Participants received 100 U/mL insulin degludec administered SC once daily (QD) over a 52-week treatment period, followed by a 5-week safety follow-up period.
Period: Treatment Period
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Started | 466 | 462
Participants Using GLP-1 Receptor Agonists | 232 | 232
Participants Not Using GLP-1 Receptor Agonists | 234 | 230
Received at Least One Dose of Study Drug | 466 | 462
Completed | 441 | 439
Not Completed | 25 | 23
Not completed — Adverse Event | 3 | 3
Not completed — Assigned treatment by mistake | 3 | 4
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 6 | 3
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol deviation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 11
Period: Follow-Up Period
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Started (Per the statistical analysis plan, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.) | 445 | 444
Completed | 441 | 439
Not Completed | 4 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol deviation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 500 U/mL - Insulin Efsitora Alfa: Participants received 500 U/mL insulin efsitora alfa administered SC QW over a 52-week treatment period, followed by a 5-week safety follow-up period.
- 100 U/mL - Insulin Degludec: Participants received 100 U/mL insulin degludec administered SC QD over a 52-week treatment period, followed by a 5-week safety follow-up period.
- Total: Total of all reporting groups
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec | Total
Number analyzed (Participants) | 466 | 462 | 928
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.6) | 57.3 (11) | 57.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 197 | 382
  Male | 281 | 265 | 546
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 123 | 242
  Not Hispanic or Latino | 345 | 335 | 680
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 34 | 36 | 70
  Asian | 163 | 164 | 327
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 27 | 58
  White | 235 | 233 | 468
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 40 | 43 | 83
  Canada | 18 | 23 | 41
  China | 67 | 67 | 134
  Czechia | 48 | 50 | 98
  Germany | 30 | 27 | 57
  Greece | 17 | 15 | 32
  Japan | 71 | 73 | 144
  Mexico | 50 | 49 | 99
  South Korea | 11 | 8 | 19
  United States | 114 | 107 | 221
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.21 (0.96) | 8.23 (0.96) | 8.22 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 52 [Noninferiority Analysis]
Description: * HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  * Least Squares (LS) mean was determined using Analysis of Covariance (ANCOVA) model with Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline or Week 52. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 463 | 458
Percentage of HbA1c | -1.26 (0.0470) | -1.17 (0.0473)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Non-Inferiority — 0.4% noninferiority margin (NIM); ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.22 to 0.04]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 52 in Participants Using GLP-1 Receptor Agonists [Noninferiority Analysis]
Description: * HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  * LS mean was determined using ANCOVA model with Baseline + Country + SU Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 52
Population: All randomized participants who continued using GLP-1 receptor agonists and received at least one dose of the study drug, had HbA1c measurement at baseline or Week 52. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 230 | 231
Percentage of HbA1c | -1.26 (0.0699) | -1.19 (0.0696)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Non-Inferiority — 0.4% noninferiority margin (NIM); ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.26 to 0.13]

3. Secondary Outcome: Change From Baseline in HbA1c at Week 52 in Participants Not Using GLP-1 Receptor Agonists [Noninferiority Analysis]
Description: as for outcome 2
Time Frame: Baseline, Week 52
Population: All randomized participants who were not using GLP-1 receptor agonists and received at least one dose of the study drug, had HbA1c measurement at baseline or Week 52. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 233 | 227
Percentage of HbA1c | -1.26 (0.0627) | -1.15 (0.0639)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Non-Inferiority — 0.4% noninferiority margin (NIM); ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.28 to 0.07]

4. Secondary Outcome: Change From Baseline in HbA1c at Week 52 [Superiority Analysis]
Description: * HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  * LS mean was determined using ANCOVA model with Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 463 | 458
Percentage of HbA1c | -1.26 (0.0470) | -1.17 (0.0473)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.188, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.22 to 0.04]

5. Secondary Outcome: Percentage of Time in the Blood Glucose Range Between 70 and 180 mg/dL [3.9 and 10.0 mmol/L] - Week 48 to Week 52
Description: * Percentage of time spent within the blood glucose range of 70 to 180 milligrams per deciliter (mg/dL) [3.9 to 10.0 millimoles per liter (mmol/L)], as measured during the continuous glucose monitoring (CGM) session over a 24-hour period, from Week 48 to Week 52.
  * LS mean was determined using ANCOVA model with Baseline + Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization + SU Use at Randomization + Treatment (Type III sum of squares) as variables. Missing data at baseline were imputed using multiple imputation under the assumption of missing at random, while missing data at Week 48-52 were imputed using a return-to-baseline multiple imputation approach.
Time Frame: Week 48 to Week 52
Population: All randomized participants who took at least 1 dose of the study drug and had CGM data collected using the Dexcom G6 system at baseline or Week 48-52 were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded. As pre-specified in the statistical analysis plan, outcome data were analyzed only from CGM data collected by the Dexcom G6 system.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 387 | 381
Percentage of time | 64.27 (1.076) | 61.18 (1.085)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.043, ANCOVA; LS Mean Difference = 3.09, 95% CI 2-sided [0.09 to 6.08]

6. Secondary Outcome: Change From Baseline in HbA1c at Week 26 [Superiority Analysis]
Description: * HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  * LS mean was determined using ANCOVA model with Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 26 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline or Week 26. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 463 | 458
Percentage of HbA1c | -1.37 (0.0394) | -1.30 (0.0397)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.260, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.17 to 0.05]

7. Secondary Outcome: Percentage of Time in the Blood Glucose Range Between 70 and 180 mg/dL [3.9 and 10.0 mmol/L] - Week 22 to Week 26
Description: * Percentage of time spent within the blood glucose range of 70 to 180 mg/dL (3.9 to 10.0 mmol/L), as measured during the CGM session over a 24-hour period, from Week 22 to Week 26.
  * LS mean was determined using ANCOVA model with Baseline + Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization + SU Use at Randomization + Treatment (Type III sum of squares) as variables. Missing data at baseline were imputed using multiple imputation under the assumption of missing at random, while missing data at Week 22-26 were imputed using a return-to-baseline multiple imputation approach.
Time Frame: Week 22 to Week 26
Population: All randomized participants who took at least 1 dose of the study drug and had CGM data collected using the Dexcom G6 system at baseline or Week 22-26 were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded. As pre-specified in the statistical analysis plan, outcome data were analyzed only from CGM data collected by the Dexcom G6 system.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 385 | 382
Percentage of time | 66.12 (0.991) | 65.85 (0.990)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.848, ANCOVA; LS Mean Difference = 0.27, 95% CI 2-sided [-2.48 to 3.02]

8. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG)
Description: Change from baseline in fasting blood glucose measured by self-monitoring blood glucose (SMBG).
Time Frame: Baseline, Week 26, Week 52
Population: All randomized participants who received at least 1 dose of the study drug and had evaluable data for this outcome at Baseline, Week 26, or Week 52 were included.For the Week 26 analysis data from Baseline and Week 26 were used and for Week 52 analysis data from Baseline and Week 52 data were used.Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter (mg/dL)
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 458 | 451
Milligram per deciliter (mg/dL)
  Week 26 | -57.86 (1.491) | -63.04 (1.500)
  Week 52: number analyzed (Participants) | 458 | 448
  Week 52 | -59.77 (1.400) | -59.97 (1.405)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 26 (Statistical Analysis) - LS mean was determined using ANCOVA model with Baseline + Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization + SU Use at Randomization + Treatment (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at week 26 were imputed by return-to-baseline multiple imputations approach; Test type: Superiority; p = 0.014, ANCOVA; LS Mean Difference = 5.18, 95% CI 2-sided [1.06 to 9.30]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 52 (Statistical Analysis) - LS mean was determined using ANCOVA model with Baseline + Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization + SU Use at Randomization + Treatment (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at week 52 were imputed by return-to-baseline multiple imputations approach; Test type: Superiority; p = 0.918, ANCOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-3.65 to 4.06]

9. Secondary Outcome: Glucose Variability
Description: * Glucose variability measured as coefficient of variation (CV) for blood glucose during the CGM session over a 24-hour period, between Week 22 to Week 26 and Week 48 to Week 52 was reported.
  * LS mean was determined using Mixed Model Repeated Measures (MMRM) model with Baseline + Country +HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 22 to Week 26 and Week 48 to Week 52
Population: All randomized participants who took at least 1 dose of the study drug and had Dexcom G6 system CGM data collected at baseline and at least 1 post-baseline value were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded. As pre-specified in the statistical analysis plan, outcome data were analyzed only from CGM data collected by the Dexcom G6 system.
Measure: Least Squares Mean (Standard Error); unit: Percentage of CV
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 368 | 360
Percentage of CV
  Week 22 to Week 26 | 26.31 (0.250) | 26.67 (0.251)
  Week 48 to Week 52 | 26.29 (0.243) | 26.81 (0.246)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 22 to Week 26 (Statistical Analysis); Test type: Superiority; p = 0.310, Mixed Models Analysis; LS Mean Difference = -0.36, 95% CI 2-sided [-1.06 to 0.34]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 48 to Week 52 (Statistical Analysis); Test type: Superiority; p = 0.138, Mixed Models Analysis; LS Mean Difference = -0.51, 95% CI 2-sided [-1.19 to 0.17]

10. Secondary Outcome: Basal Insulin Dose
Description: * The insulin dose was calculated based on the participant's entry of daily or weekly insulin doses in an electronic diary. The average weekly basal insulin dose at Week 26 and Week 52 was reported.
  * LS mean was determined using MMRM model with Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 26 and Week 52
Population: All randomized participants who received at least one dose of the study drug and had a baseline and at least one post-baseline value for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Units per week (U/week)
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 463 | 457
Units per week (U/week)
  Week 26 | 292.8 (6.30) | 305.9 (6.17)
  Week 52 | 314.7 (6.25) | 334.4 (6.22)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 26 (Statistical Analysis); Test type: Superiority; p = 0.136, Mixed Models Analysis; LS Mean Difference = -13.2, 95% CI 2-sided [-30.5 to 4.1]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 52 (Statistical Analysis); Test type: Superiority; p = 0.026, Mixed Models Analysis; LS Mean Difference = -19.7, 95% CI 2-sided [-37.0 to -2.4]

11. Secondary Outcome: Hypoglycemia Event Rate
Description: * A hypoglycemic event with blood glucose (BG) levels of less than (<) 54 mg/dL (3.0 mmol/L) [Level 2] or Severe Hypoglycemia [Level 3] was reported. A severe hypoglycemic event was characterized by altered mental or physical status, requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia.
  * Group mean was reported and determined by Negative binomial model using Number of episodes = HbA1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Error); unit: Events per participant-year of exposure
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 466 | 462
Events per participant-year of exposure | 0.58 (0.062) | 0.45 (0.058)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.111, Negative binomial model; Relative Rate = 1.30, 95% CI 2-sided [0.94 to 1.78]

12. Secondary Outcome: Nocturnal Hypoglycemia Event Rate
Description: * The event rate of participant-reported clinically significant nocturnal hypoglycemia (defined as blood glucose level <54 mg/dL (3.0 mmol/L) or severe hypoglycemia and occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment phase up to week 52.
  * Group mean was reported and determined by Negative binomial model using Number of episodes = HbA1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Error); unit: Events per participant-year of exposure
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 466 | 462
Events per participant-year of exposure | 0.08 (0.018) | 0.08 (0.018)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Test type: Superiority; p = 0.983, Negative binomial model; Relative Rate = 1.01, 95% CI 2-sided [0.53 to 1.89]

13. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported. LS mean was determined by MMRM model with Baseline + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26, Week 52
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post- baseline value for this outcome were included.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 465 | 461
Kilogram (kg)
  Week 26 | 3.16 (0.158) | 2.66 (0.158)
  Week 52 | 3.60 (0.158) | 3.54 (0.159)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 26 (Statistical Analysis); Test type: Superiority; p = 0.025, Mixed Models Analysis; LS Mean Difference = 0.50, 95% CI 2-sided [0.064 to 0.94]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 52 (Statistical Analysis); Test type: Superiority; p = 0.801, Mixed Models Analysis; LS Mean Difference = 0.056, 95% CI 2-sided [-0.38 to 0.50]

14. Secondary Outcome: Percentage of Time in Hypoglycemia Range With Blood Glucose <70 mg/dL (3.9 mmol/L)
Description: * Percentage of time spent in the hypoglycemia range with blood glucose <70 mg/dL (3.9 mmol/L), as measured during the CGM session over a 24-hour period from Week 8 to Week 12, Week 22 to Week 26, and Week 48 to Week 52 was reported.
  * LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 8 to Week 12, Week 22 to Week 26 and Week 48 to Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 368 | 360
Percentage of time
  Week 8 to Week 12 | 1.06 (0.101) | 0.93 (0.103)
  Week 22 to Week 26 | 1.55 (0.137) | 1.25 (0.137)
  Week 48 to Week 52 | 1.49 (0.150) | 1.19 (0.152)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 8 to Week 12 (Statistical Analysis); Test type: Superiority; p = 0.374, Mixed Models Analysis; LS Mean Difference = 0.13, 95% CI 2-sided [-0.15 to 0.41]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 22 to Week 26 (Statistical Analysis); Test type: Superiority; p = 0.130, Mixed Models Analysis; LS Mean Difference = 0.29, 95% CI 2-sided [-0.09 to 0.67]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 48 to Week 52 (Statistical Analysis); Test type: Superiority; p = 0.162, Mixed Models Analysis; LS Mean Difference = 0.30, 95% CI 2-sided [-0.12 to 0.72]

15. Secondary Outcome: Percentage of Time in Hypoglycemia Range With Blood Glucose <54 mg/dL (3.0 mmol/L)
Description: * Percentage of time spent in the hypoglycemia range with blood glucose < 54 mg/dL (3.0 mmol/L), as measured during the CGM session over a 24-hour period from Week 8 to Week 12, Week 22 to Week 26, and Week 48 to Week 52, was reported.
  * LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 8 to Week 12, Week 22 to Week 26 and Week 48 to Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 368 | 360
Percentage of time
  Week 8 to Week 12 | 0.24 (0.041) | 0.27 (0.041)
  Week 22 to Week 26 | 0.33 (0.037) | 0.28 (0.037)
  Week 48 to Week 52 | 0.32 (0.043) | 0.30 (0.043)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 8 to Week 12 (Statistical Analysis); Test type: Superiority; p = 0.594, Mixed Models Analysis; LS Mean Difference = -0.03, 95% CI 2-sided [-0.15 to 0.08]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 22 to Week 26 (Statistical Analysis); Test type: Superiority; p = 0.266, Mixed Models Analysis; LS Mean Difference = 0.06, 95% CI 2-sided [-0.04 to 0.16]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 48 to Week 52 (Statistical Analysis); Test type: Superiority; p = 0.791, Mixed Models Analysis; LS Mean Difference = 0.02, 95% CI 2-sided [-0.10 to 0.14]

16. Secondary Outcome: Percentage of Time in Hyperglycemia Range With Blood Glucose >180 mg/dL (10.0 mmol/L)
Description: * Percentage of time spent in the hyperglycemia range with blood glucose greater than (>) 180 mg/dL (10.0 mmol/L), as measured during the CGM session over a 24-hour period from Week 8 to Week 12, Week 22 to Week 26, and Week 48 to Week 52 was reported.
  * LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 8 to Week 12, Week 22 to Week 26 and Week 48 to Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 368 | 360
Percentage of time
  Week 8 to Week 12 | 31.99 (0.925) | 32.40 (0.939)
  Week 22 to Week 26 | 28.93 (0.999) | 29.87 (1.007)
  Week 48 to Week 52 | 29.66 (1.074) | 33.05 (1.086)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 8 to Week 12 (Statistical Analysis); Test type: Superiority; p = 0.757, Mixed Models Analysis; LS Mean Difference = -0.41, 95% CI 2-sided [-3.00 to 2.18]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 22 to Week 26 (Statistical Analysis); Test type: Superiority; p = 0.511, Mixed Models Analysis; LS Mean Difference = -0.93, 95% CI 2-sided [-3.72 to 1.85]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 48 to Week 52 (Statistical Analysis); Test type: Superiority; p = 0.027, Mixed Models Analysis; LS Mean Difference = -3.39, 95% CI 2-sided [-6.39 to -0.39]

17. Secondary Outcome: Change From Baseline in Treatment-Related Impact Measures for Diabetes (TRIM-D) -Total Score at Week 26 and Week 52
Description: * The TRIM-D is a participant-reported measure designed to assess the impact of diabetes treatment on individuals' functioning and well-being across different diabetes treatments. The questionnaire includes 28 items grouped into 5 sub-domains: treatment burden, daily life, diabetes management, compliance, and psychological health. Each item is assessed on a 5-point scale, with higher scores indicating better health status. All items were summed to obtain a total raw score, which was transformed to a scale of 0 to 100 to obtain a total score. The total score range is 0-100, with a higher total score indicating better overall health and well-being, while a lower total score indicates worse health or well-being.
  * LS mean was determined using MMRM model with Baseline + Country + HbA1c Stratum at Baseline + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26, Week 52
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post- baseline value for this outcome.Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 444 | 445
score on a scale
  Week 26 | 8.84 (0.507) | 7.18 (0.507)
  Week 52 | 8.82 (0.519) | 6.81 (0.517)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 26 (Statistical Analysis); Test type: Superiority; p = 0.021, Mixed Models Analysis; LS Mean Difference = 1.66, 95% CI 2-sided [0.26 to 3.07]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Week 52 (Statistical Analysis); Test type: Superiority; p = 0.006, Mixed Models Analysis; LS Mean Difference = 2.00, 95% CI 2-sided [0.57 to 3.44]

18. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey Version 2 (SF-36v2) Acute Form (Physical-Component and Mental-Component) Scores at Week 26 and Week 52
Description: The SF-36v2 is a participant-reported measure designed to assess health status using 36 items across 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Each domain is scored individually, and information from these 8 domains is further aggregated into 2 health component summary scores, the Physical Component Summary and Mental Component Summary. Scoring of each domain and both summary scores are norm based and presented in the form of T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate better levels of function and/or better health. Range cannot be specified in norm-based scores.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 431 | 434
T-score
  Physical Component Score at Week 26 | 0.29 (0.344) | 0.49 (0.345)
  Mental Component Score at Week 26 | 0.018 (0.380) | 0.34 (0.381)
  Physical Component Score at Week 52 | 0.027 (0.349) | -0.14 (0.351)
  Mental Component Score at Week 52 | 0.014 (0.386) | 0.25 (0.389)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Physical Component Score at Week 26 (Statistical Analysis) -LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.638, Mixed Models Analysis; LS Mean Difference = -0.20, 95% CI 2-sided [-1.03 to 0.63]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Mental Component Score at Week 26 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.499, Mixed Models Analysis; LS Mean Difference = -0.32, 95% CI 2-sided [-1.24 to 0.60]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Physical Component Score at Week 52 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.695, Mixed Models Analysis; LS Mean Difference = 0.17, 95% CI 2-sided [-0.68 to 1.01]
Statistical Analysis 4: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; Mental Component Score at Week 52 (Statistical Analysis) -LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use at Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.626, Mixed Models Analysis; LS Mean Difference = -0.23, 95% CI 2-sided [-1.17 to 0.71]

19. Secondary Outcome: Change From Baseline in EuroQuality of Life (EuroQol) - 5 Dimensions-5 Levels (EQ-5D-5L) Health State Index and EQ Visual Analog Scale (VAS) Scores at Week 26 and Week 52
Description: The EQ-5D-5L is a multidimensional, health-related, quality-of-life instrument. It includes 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that are assessed at 5 levels of response (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). The scores in the 5 dimensions were summarized into a health state index score. A single health-state index value was derived, which ranges from less than 0 (health state equivalent to death, negative values are valued as worse than death) to 1 (perfect health). The EQ VAS rates the participants' perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health). This score provides a composite picture of the respondent's health status.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
Number analyzed (Participants) | 430 | 434
Score on a scale
  EQ-5D-5L Health State Index Score at Week 26 | -0.018 (0.0078) | -0.004 (0.0078)
  EQ VAS Score at Week 26 | 1.07 (0.701) | 2.18 (0.699)
  EQ-5D-5L Health State Index Score at Week 52 | -0.018 (0.0077) | -0.008 (0.0077)
  EQ VAS Score at Week 52 | 1.56 (0.733) | 1.91 (0.739)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; EQ-5D-5L Health State Index Score at Week 26 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.128, Mixed Models Analysis; LS Mean Difference = -0.015, 95% CI 2-sided [-0.034 to 0.004]
Statistical Analysis 2: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; EQ VAS Score at Week 26 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.196, Mixed Models Analysis; LS Mean Difference = -1.11, 95% CI 2-sided [-2.80 to 0.58]
Statistical Analysis 3: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; EQ-5D-5L Health State Index Score at Week 52 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.285, Mixed Models Analysis; LS Mean Difference = -0.010, 95% CI 2-sided [-0.029 to 0.008]
Statistical Analysis 4: Comparison: 500 U/mL - Insulin Efsitora Alfa vs 100 U/mL - Insulin Degludec; EQ VAS Score at Week 52 (Statistical Analysis) - LS mean was determined using MMRM model with Baseline + HbA1c Stratum at Baseline + Country + GLP-1 RA Use Randomization Flag + SU Use at Randomization Flag + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.701, Mixed Models Analysis; LS Mean Difference = -0.35, 95% CI 2-sided [-2.15 to 1.44]

ADVERSE EVENTS:
Time Frame: Baseline to end of follow-up (up to 57 weeks)
Description: * All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received.
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 500 U/mL - Insulin Efsitora Alfa | 100 U/mL - Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 2/466 | 1/462
Serious Adverse Events (participants affected / at risk) | 41/466 | 38/462
Other Adverse Events (participants affected / at risk) | 195/466 | 224/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora Alfa (N=466) | 100 U/mL - Insulin Degludec (N=462)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal ischaemia (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign spleen tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1/185 (1) | 0/197 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/281 (1) | 0/265 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/185 (1) | 0/197 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora Alfa (N=466) | 100 U/mL - Insulin Degludec (N=462)
Diarrhoea (Gastrointestinal disorders) | 31 (36) | 32 (48)
Nausea (Gastrointestinal disorders) | 26 (27) | 26 (29)
Covid-19 (Infections and infestations) | 37 (38) | 51 (51)
Influenza (Infections and infestations) | 18 (22) | 26 (31)
Nasopharyngitis (Infections and infestations) | 43 (50) | 41 (50)
Upper respiratory tract infection (Infections and infestations) | 37 (52) | 46 (63)
Urinary tract infection (Infections and infestations) | 17 (20) | 29 (35)
Drug titration error (Injury, poisoning and procedural complications) | 33 (58) | 55 (86)
Weight increased (Investigations) | 28 (30) | 20 (20)
Headache (Nervous system disorders) | 21 (30) | 28 (47)

LIMITATIONS AND CAVEATS:
As prespecified in the statistical analysis plan, outcome analyses related to Continuous Glucose Monitoring (CGM) were conducted using data from the Dexcom G6 system, which was used at all study sites except those in China. In China, CGM data were collected using the Libre FreeStyle H system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05362058/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT05362058/SAP_001.pdf